CLINICAL TRIAL: NCT06999759
Title: Concealment of Chemotherapy Drug Serum With a Picture Box Effect on Anxiety, Nausea and Vomiting in Children: A Prospective Randomized Controlled Study
Brief Title: Concealment of Chemotherapy Drug Serum With a Picture Box Effect on Anxiety, Nausea and Vomiting in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Associate Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/10-03
Record Dates: First submitted 2025-05-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Nursing Caries; Art Therapy
Keywords: Chemotherapy; Chemotherapy drug serum; Child; Anxiety; Nausea and Vomiting
MeSH Terms: conditions — Anxiety Disorders; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of cute serum boxes (Experimental): Children in the study group were provided with cute picture boxes with their own pictures hanging on them to receive chemotherapy.
  Interventions: Device: cute serum box; Other: coloring book and coloring pencils
- Control Group (No Intervention): The chemotherapy drug serum of the children in the control group was not concealed by the designed picture box, and they continued their treatment routinely.

INTERVENTIONS:
Device: cute serum box — After the children in the intervention group were made to draw pictures, they were glued to the designed cute serum box and chemotherapy drug serum was hidden and they were provided to receive their treatment.
  Arms: group of cute serum boxes
Other: coloring book and coloring pencils — Children in the intervention group were provided with a coloring book and coloring pencils to make a picture to hang on the picture box.
  Arms: group of cute serum boxes

SUMMARY:
The aim of this study was to present the results of the effect of concealing chemotherapy drug serum with a picture box on children's anxiety, nausea and vomiting. The study was planned with children aged 5-10 years who met the inclusion criteria.

In this randomised controlled study, 70 children with cancer who are hospitalised in Marmara University Hospital and meet the inclusion criteria will be divided into two equal groups. The first group (intervention group) receives chemotherapy in chemotherapy boxes in which pictures made by the children are pasted before starting chemotherapy. In the second group (control group), children do not draw and chemotherapy boxes are not used. In both groups, the'' Child Anxiety Scale - State Anxiety Scale'' and the' Nausea - Vomiting Thermometer Scale in Children with Cancer'' will be used to assess children's state anxiety and nausea and vomiting. The scores given by the children will be noted by the researcher and the observer 5 minutes before the treatment and immediately after the end of the treatment in the scale scores section of the 'Child monitoring and evaluation form during chemotherapy'.

DETAILED DESCRIPTION:
Childhood cancers require intensive health care and have a high burden of disease. Childhood cancers have turned into a chronic disease that causes increasing physical and psychosocial symptoms all over the world and in our country, rather than a fatal disease, due to developments in multi-agent chemotherapy protocols, the use of targeted chemotherapeutic agents, intrathecal applications and supportive care.

Chemotherapy is accepted as the main treatment in childhood cancers. Symptoms related to chemotherapy in children diagnosed with cancer affect the continuity of treatment, life expectancy, morbidity, mortality and quality of life of the child.

In the literature review, studies on anxiety, depression and behavioural changes in the first year after diagnosis reported that anxiety was an important problem after diagnosis and the number of children scoring in the at-risk/clinical range of depression was high.

Nausea and vomiting is one of the most common symptoms in the treatment of childhood cancers. In studies, 60.9% of children receiving inpatient chemotherapy had nausea within one week after treatment. In a study on the presence, severity, risk factors and the effect on quality of life of symptoms related to nausea and vomiting in children with cancer in the first year of treatment, 41.8% and 42.9% of patients experienced nausea in the 3rd and 6th month after diagnosis, respectively.

İn the literature review, no study was found to reduce anxiety, nausea and vomiting symptoms of children diagnosed with cancer by using art therapy together with cognitive method during chemotherapy by taking into account the smell, appearance and previous negative experiences of chemotherapy serum drug.

In conclusion, cancer diagnosis, invasive interventions, long-term hospitalisation, long-term procedures, protocols and chemotherapy have negative effects on children.In this study, the effects of concealment of the drug serum during intravenous chemotherapy on anxiety, nausea and vomiting of children aged 5-10 years who are receiving chemotherapy for cancer will be compared. Art therapy, which is one of the therapeutic approaches during treatment, is aimed to improve the treatment process by diverting the child's attention and to change the negative feelings and thoughts caused by the smell, appearance, previous experiences of chemotherapy serum drug.

ELIGIBILITY:
Inclusion Criteria:

* 5-10 years old (The scale used is between this age group, these children should be willing to draw and should be suitable for their developmental periods)
* Inpatients with cancer,
* Those receiving the second and subsequent courses of chemotherapy,
* Previous chemotherapy experience,
* Those receiving chemotherapy drugs, the duration of chemotherapy lasting an average of 1 to 6 hours
* Those taking chemotherapy drugs with minimal, low and moderate severity of nausea and vomiting,
* Children whose parents agreed to participate in the study were included in the study.

Exclusion Criteria:

* Those in the last stage of cancer (experiencing the side effects of treatment intensively during hospitalisation due to the disease and symptoms causing complications)
* Those receiving oral chemotherapy,
* Those who experience intense side effects of chemotherapy (febrile neutropenia, bleeding, allergic reactions),
* People with mental problems (depression, anxiety disorders, disruptive behaviour disorders, neurodevelopmental disorders),
* People on antidepressant medication,
* Those who have a physical disability (e.g. amputation, lack/inability to use arms, hands and fingers, visual or hearing impairment, etc.) to paint during chemotherapy, and
* Children taking medicines with high severity of nausea and vomiting were not included in the study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
. The change in child anxiety scale state scale (CAS-D) scores of the group receiving chemotherapy drug serum with picture box | 5 minutes before the start of chemotherapy medication and immediately after the end of treatment.]
  It was determined 5 minutes before the planned therapeutic process and immediately after the end of the treatment with the ''Child Anxiety Scale-Situation Scale''.An increase in the scale score indicates an increase in the child's anxiety. The total score varies between 0-10 points.The lowest score that can be selected from the scale is ''0'' and the highest score is ''10''.

SECONDARY OUTCOMES:
Change in nausea-vomiting thermometer scale (NVT) scores of the group receiving chemotherapy drug serum with picture box. | 5 minutes before the start of chemotherapy medication and immediately after the end of treatment.
  The severity of nausea and vomiting was determined with the "Nausea-Vomiting Thermometer Scale in Children with Cancer" 5 minutes before the planned therapeutic process and immediately after the end of the treatment. An increase in the scale score indicates that the child's complaint of nausea and vomiting increased. The total score range varies between 1 and 5 points. The lowest score that can be selected from the scale is '1' and the highest score is '5'.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem ERGÜN, Principal Investigator — Maltepe University School of Nursing İstanbul,Turkey
Locations (1):
- Marmara Unıvesıty Educatıon And Research Hospıtal Istanbul, Pendik, Turkey, 34000 ., Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Saeidzadeh S, Kamalumpundi V, Chi NC, Nair R, Gilbertson-White S. Web and mobile-based symptom management interventions for physical symptoms of people with advanced cancer: A systematic review and meta-analysis. Palliat Med. 2021 Jun;35(6):1020-1038. doi: 10.1177/02692163211006317. Epub 2021 Apr 12. PMID 33840271
- [Background] Çavuşoğlu, H. (2019). Çocuk Sağlığı Hemşireliği. Cilt 2, Ankara: Sistem Ofset Matbaacılık.
- [Background] Withycombe JS, Haugen M, Zupanec S, Macpherson CF, Landier W. Consensus Recommendations From the Children's Oncology Group Nursing Discipline's State of the Science Symposium: Symptom Assessment During Childhood Cancer Treatment. J Pediatr Oncol Nurs. 2019 Jul/Aug;36(4):294-299. doi: 10.1177/1043454219854983. PMID 31307318
- [Background] Ward ZJ, Yeh JM, Bhakta N, Frazier AL, Atun R. Estimating the total incidence of global childhood cancer: a simulation-based analysis. Lancet Oncol. 2019 Apr;20(4):483-493. doi: 10.1016/S1470-2045(18)30909-4. Epub 2019 Feb 26. PMID 30824204
- [Background] Tripathi, A. K., David, A., Govil, T., Rauniyar, S., Rathinam, N. Κ., Goh, K. M., Sani, R. K. (2020). Environmental Remediation of Antineoplastic Drugs: Present Status, Challenges, and Future Directions. Processes, 8(7), 747. doi:10.3390/pr8070747.
- [Background] Nie Y, Tian Y, Han X. Music Nursing as Complementary Therapy Improves Anxiety, Fatigue, and Quality of Life in Children with Acute Leukaemia: A Retrospective Study. Noise Health. 2024 Jan-Mar 01;26(120):25-29. doi: 10.4103/nah.nah_33_24. Epub 2024 Mar 23. PMID 38570307
- [Background] Myers RM, Balsamo L, Lu X, Devidas M, Hunger SP, Carroll WL, Winick NJ, Maloney KW, Kadan-Lottick NS. A prospective study of anxiety, depression, and behavioral changes in the first year after a diagnosis of childhood acute lymphoblastic leukemia: a report from the Children's Oncology Group. Cancer. 2014 May 1;120(9):1417-25. doi: 10.1002/cncr.28578. Epub 2014 Jan 28. PMID 24473774
- [Background] Hu H, Shear D, Thakkar R, Thompson-Lastad A, Pinderhughes H, Hecht FM, Lown EA. Acupressure and Therapeutic Touch in Childhood Cancer to Promote Subjective and Intersubjective Experiences of Well-being During Curative Treatment. Glob Adv Health Med. 2019 Sep 30;8:2164956119880143. doi: 10.1177/2164956119880143. eCollection 2019. PMID 31632842
- [Background] Braam KI, van Dijk-Lokkart EM, Kaspers GJL, Takken T, Huisman J, Buffart LM, Bierings MB, Merks JHM, van den Heuvel-Eibrink MM, Veening MA, van Dulmen-den Broeder E. Effects of a combined physical and psychosocial training for children with cancer: a randomized controlled trial. BMC Cancer. 2018 Dec 27;18(1):1289. doi: 10.1186/s12885-018-5181-0. PMID 30587148
- [Background] Gerçeker, G. Ö., Ayar, D., Özdemir, Z., ve Bektaş, M. (2018). Çocuk Anksiyete Skalası-Durumluluk ve Çocuk Korku Ölçeğinin Türk Diline Kazandırılması. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 11(1), 9-13.
- [Background] Akdeniz Kudubes A, Bektas M. Developing the Nausea and Vomiting Thermometer Scale in children with cancer. Turk J Med Sci. 2022 Feb;52(1):166-174. doi: 10.3906/sag-2005-88. Epub 2022 Feb 22. PMID 34544217
- [Background] Altay N, Kilicarslan-Toruner E, Sari C. The effect of drawing and writing technique on the anxiety level of children undergoing cancer treatment. Eur J Oncol Nurs. 2017 Jun;28:1-6. doi: 10.1016/j.ejon.2017.02.007. Epub 2017 Mar 2. PMID 28478846
- [Background] Aguilar BA. The Efficacy of Art Therapy in Pediatric Oncology Patients: An Integrative Literature Review. J Pediatr Nurs. 2017 Sep-Oct;36:173-178. doi: 10.1016/j.pedn.2017.06.015. Epub 2017 Jun 30. PMID 28888499